CLINICAL TRIAL: NCT04095949
Title: Absorption, Metabolism and Excretion of Artichoke Polyphenols in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Lecturer in Nutrition, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Artichoke Study
Record Dates: First submitted 2019-07-24; First posted 2019-09-19 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Healthy Men and Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artichokes (Experimental): 1 day of artichokes intake
  Interventions: Dietary Supplement: Artichokes

INTERVENTIONS:
Dietary Supplement: Artichokes — Approximately 200 g of cooked artichokes

SUMMARY:
A number of studies have reported the presence of polyphenolic compounds in artichokes, being the most abundant the caffeoylquinic acids (CQAs), which are esters between quinic acid and the hydroxycinnamate caffeic acid. The fate of artichoke polyphenols in humans after ingestion is currently unknown. The acute study will provide novel information on the bioavailability and metabolism of artichoke polyphenols, which will give important insights to understand the potential health benefits of artichoke consumption.

Health men and women participants (n=8) aged between 18 to 40 years old will be recruited. Participants will consume a normal ration of artichokes once. The participants will provide the investigators with urine and blood samples for polyphenol analysis at baseline and at different time points until 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women aged 18-40 years old
2. Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
3. Are able to understand the nature of the study
4. Able to give signed written informed consent
5. Signed informed consent form

Exclusion Criteria:

1. Metabolic disease
2. Chronic disease or medications
3. BMI not between 18.5 and 30
4. Allergies to artichokes or other significant food allergy.
5. Subjects under medication or on vitamin/dietary supplements.
6. Subjects who reported participant in another study within one month before the study start
7. Pregnant woman or planning to become pregnant in the next month
8. Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change in qualitative identification of polyphenols and their metabolites of artichokes in plasma between baseline and 24h post consumption | Baseline, 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours and 24 hours
  Change in polyphenols and their metabolites in plasma between baseline and 24h post consumption will be measured by identifying qualitatively metabolites from artichokes at different time points using chromatography coupled with mass spectrometry analytical techniques (UPLC-MS).
Change in qualitative identification of polyphenols and their metabolites of artichokes in urine between baseline and 24h post consumption | Baseline, 0-2 hours, 2-4 hours, 4-8 hours and 8-24 hours
  Change in polyphenols and their metabolites in urine between baseline and 24h post consumption will be measured by identifying qualitatively metabolites from artichokes at different time points using chromatography coupled with mass spectrometry analytical techniques (UPLC-MS).
Change in the plasmatic concentration of polyphenols (nanomol/L) and their metabolites of artichokes between baseline and 24h post consumption | Baseline, 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours and 24 hours
  Bioavailability and metabolism from artichoke polyphenols will be studied by evaluating changes in artichoke polyphenols concentration (nanomol/L) in plasma samples at different time points using chromatography coupled with mass spectrometry analytical techniques (UPLC-MS).
Change in the concentration of polyphenols in urine (nanomol/L) and their metabolites of artichokes between baseline and 24h post consumption | Baseline, 0-2 hours, 2-4 hours, 4-8 hours and 8-24 hours
  Metabolism and excretion from artichoke polyphenols will be studied by evaluating changes in artichoke polyphenols concentration (nanomol/L) in urine samples at different time points using chromatography coupled with mass spectrometry analytical techniques (UPLC-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — ana.rodriguez-mateos@kcl.ac.uk
Locations (1):
- King's College London, Department of Nutritional Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No